CLINICAL TRIAL: NCT00726258
Title: Association of Intravenous Ketamine With Thoracic Epidural Analgesia: Effects on Pain and Respiratory Function Following Thoracotomy.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-00336-20; 2007-04
Record Dates: First submitted 2008-07-30; First posted 2008-07-31 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Thoracotomy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Drip of physiological serum
  Interventions: Drug: placebo
- 2 (Active Comparator): Drip of ketamine
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — ketamine with various concentrations
  Arms: 2
Drug: placebo — physiological serum
  Arms: 1

SUMMARY:
Thoracotomy for lung resection is deemed painful. Ketamine is now a renewed interest in preventing acute postoperative pain. A previous study performed in the service testing the association ketamine/morphine versus morphine PCA, postoperative, for patients who do not benefit from postoperative epidural thoracic surgery, has demonstrated a reduction of postoperative pain associated with a reduction of nocturnal arterial desaturation following surgery when ketamine was added to morphine.

DETAILED DESCRIPTION:
In this prospective double blind randomized study, intravenous administration of an analgesic dose of ketamine was started since the induction of general anesthesia and continued during the first 48 postoperative hours in association with epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Subject between 18 and 85 years
* subject of both sexes
* subject operated in the service of thoracic surgery of a lobectomy by thoracotomie lateral or postlaterale subject
* subject operated in settled surgery

Exclusion Criteria:

* Against indication in the epidural insanity,
* confusionnel, patient psychotic
* treatment in the long price by medicine which can interfere on the pain (morphine, antidepressants, psychotropic treatment)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To estimate the immediate postoperative analgesic effect of the association ketamine IV-thoracic epidural with regard to the use of the only epidural | 24 months

SECONDARY OUTCOMES:
To estimate the effect of the association ketamine IV thoracic epidural on the postoperative pain postponed in 1, 3 and 6 months | 24 months
To estimate the effect of the association ketamine IV thoracic epidural on the incidence of the urinary side effects and hémodynamiques of the epidural | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Françoise GAILLAT, MD, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Service de chirurgie Orthopédique-Traumatologie - Hopital Sainte Marguerite, Marseille, France

REFERENCES:
- [Derived] Joseph C, Gaillat F, Duponq R, Lieven R, Baumstarck K, Thomas P, Penot-Ragon C, Kerbaul F. Is there any benefit to adding intravenous ketamine to patient-controlled epidural analgesia after thoracic surgery? A randomized double-blind study. Eur J Cardiothorac Surg. 2012 Oct;42(4):e58-65. doi: 10.1093/ejcts/ezs398. Epub 2012 Jul 12. PMID 22790008